CLINICAL TRIAL: NCT04605822
Title: Clinical Performance of the New Artificial-intelligence Powered 3D Total Body Photography System VECTRA® in Early Melanoma Detection and Its Impact on Patients' Burden of Disease: A Prospective Cohort Study in a Real-world Setting
Brief Title: Melanoma Detection in Switzerland With VECTRA
Acronym: MELVEC
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02482; sp20Maul
Record Dates: First submitted 2020-10-21; First posted 2020-10-28 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Melanoma (Skin)
Keywords: 3D total body photography (TBP); 2D sequential digital dermatoscopic imaging (SDDI); skin malignancy; artificial intelligence (AI)- based tools; 3D TBP Vectra® WB360 system; FotoFinder ATBM® Master; SkinVision®
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 3D imaging Total Body Photography Vectra® WB360 — 3D Total Body Photography Vectra® WB360 (Canfield Scientific, Parsippany, New Jersey, USA) and its digital dermoscopic camera (VISIOMED® D200evo dermatoscope) and scoring of pigmented skin lesions. All participants of this study will undergo 3D TBP at baseline and the follow-up visits up to month 24.
Device: 2D imaging FotoFinder ATBM® Master imaging system — 2D imaging with FotoFinder® Mole Analyzer and scoring of pigmented skin lesions. All participants of this study will undergo 2D imaging FotoFinder ATBM® Master imaging system at baseline and the follow-up visits up to month 24.
Device: Smartphone application (SkinVision®) — Smartphone application for all dermatoscopically documented pigmented skin lesions in all study participations and record of risk assessment of the health application (low, medium or high risk) to compare the app's accuracy in risk assessment with the AI tools and the dermatologist. The SkinVision® smartphone app is CE certified.of skin lesions. All participants of this study will undergo Smartphone application (SkinVision®) at baseline and the follow-up visits up to month 12.
Other: Standard-of-care clinical assessment of the skin — Clinical skin examination with dermatoscope by an experienced dermatologist and risk assessment of pigmented lesions (melanoma vs. naevus). All participants of this study will undergo Standard-of-care clinical assessment of the skin at baseline and the follow-up visits up to month 24.

SUMMARY:
This study is to compare 2D- and 3D-imaging and routine clinical care in early melanoma detection in a prospective large-scale real-world data set.

DETAILED DESCRIPTION:
This study is to compare the accuracy of combining human and artificial intelligence with its independent application in early melanoma detection. The Artificial Intelligence (AI)-powered 3D Total Body Photography (TBP) Vectra® WB360 system's utility and clinical performance in detecting melanoma in the real-world setting will be compared to the gold standard with clinical assessments by experienced dermatologists, to currently widespread used 2D imaging tools (FotoFinder ATBM® Master) and to the Smartphone-based algorithm application (e.g. SkinVision®). Here included are specific questions regarding the patients' subjective experience, acceptance and evaluation of modern technological examination.

Additionally, the overall psychological burden and worry of melanoma risk or disease, anxiety, depression will be compared in different groups of patients and psychological support need and real uptake of support and its predictors will be investigated in all participants.

To validate the MELVEC (Melanoma Detection in Switzerland with Vectra®) test procedure, an analysis of the measurement repeatability of computer-guided risk assessment scores for early melanoma detection will be performed. A potential benefit of this validation analysis is the optimization of study procedure for future follow-up visits and further enrolled patients in the MELVEC study. Additionally, results will shed light on the reliability of the convolutional neural networks (CNNs) investigated and help formulate recommendations for their current use. Furthermore, results will provide important data for the manufacturers regarding the systems' reliability in clinical application to help future improvement of the respective algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient
* Sufficient fluency in German language skills to complete all questionnaires of the study without external assistance
* High-risk criteria for melanoma. For "high risk" one of the following criteria needs to be fulfilled:

  * At least one previous melanoma (including melanoma in situ)
  * A diagnosis of ≥ 100 nevi
  * A diagnosis of ≥ 5 atypical nevi
  * A diagnosis of dysplastic nevus syndrome or known CDKN2A mutation
  * A strong family history (≥ 1 first- and/or second-degree relatives)

Exclusion Criteria:

* Lack of informed consent for study participation.
* Fitzpatrick skin type V-VI.
* Acute psychiatric illness or acute crisis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during melanoma consultations and the consultation in the outpatient clinic at the Department of Dermatology at the University Hospital Basel from Q4/2020 until Q4/2021.
Sampling Method: Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Analyses of histopathology reports of all excised suspectable lesions | up to 24 months
  The primary outcome, the sensitivity of human and artificial intelligence in detecting melanoma, will be measured at every study visit in case of a suspected melanoma by analysing histopathology reports of all excised suspectable lesions. The diagnosis of melanoma will be confirmed by histology. The biopsied pigmented skin lesions will be categorized as benign (melanocytic nevi / dysplastic nevi) or malignant (melanoma).
Analyses of dermatologists' assessment of each pigmented skin lesion as benign (melanocytic nevi / dysplastic nevi) or malignant (melanoma) before and after (without and with knowledge of) computer-guided risk assessment scores | up to 24 months
  Analyses of dermatologists' assessment of each pigmented skin lesion as benign (melanocytic nevi / dysplastic nevi) or malignant (melanoma) before and after computer-guided risk assessment scores by Vectra® WB360 and FotoFinder® Mole Analyzer and smartphone app.
Analyses of 2D FotoFinder® Mole Analyzer scoring of pigmented skin lesions (0.0 - 1.0) | up to 24 months
  The primary outcome, the sensitivity of human and artificial intelligence in detecting melanoma, will be measured at every study visit in case of a suspected melanoma by 2D FotoFinder® Mole Analyzer scoring of pigmented skin lesions (0.0 - 1.0). Scores 0.0 - 1.0; 0 indicating no suspicion for melanoma, 1 indicating a high suspicion for melanoma).
Analyses of 3D Vectra® WB360 imaging scoring of pigmented skin lesions (0- 10) | up to 24 months
  The primary outcome, the sensitivity of human and artificial intelligence in detecting melanoma, will be measured at every study visit in case of a suspected melanoma by analysing 3D Vectra® WB360 imaging scoring of pigmented skin lesions (0- 10). Score 0 - 10; 0 indicating no suspicion for melanoma, 10 indicating a high suspicion for melanoma).
Analyses of Smartphone app Skin Vision® scoring of pigmented skin lesions (low, medium or high risk) | up to 12 months
  The primary outcome, the sensitivity of human and artificial intelligence in detecting melanoma, will be measured at every study visit in case of a suspected melanoma by analysing Smartphone app Skin Vision® scoring of pigmented skin lesions (low, medium or high risk).

SECONDARY OUTCOMES:
Change in Distress thermometer (Patient-reported outcome) | up to 24 months
  Distress thermometer on a scale from 0-10 to address psychological distress: German version of the NCCN Distress Thermometer is used with Problem List (PL) as the screening tool for self-reported psychosocial distress, and to identify the causes of expressed distress.
Change in FACIT G7 Functional Assessment of Cancer Therapy - General - (7 item version). | up to 24 months
  The FACIT Measurement System is a collection of QOL questionnaires targeted to the management of chronic illness.
Change in Hospital Anxiety and Depression Scale (HADS) | up to 24 months
  The HADS is a 14-item self-administered questionnaire widely used to detect anxiety and depression in physically ill patients and is validated for the German language. The questionnaire has two subscales (anxiety and depression) with seven items each and a total score for each subscale (values from 0-21). Subscale scores between 0-7 indicate normal anxiety and depression levels, scores between 8-10 indicate borderline levels of anxiety and depression, and scores between 11-21 indicate clinical levels of anxiety or depression
Change in Melanoma Worry Scale (MWS) | up to 24 months
  MWS comprises four items, score 1 to 4, with possible scores ranging from 4 to 17, a higher score indicating higher levels of worry
Change in support need and uptake | up to 24 months
  Support need and uptake will be collected by questions regarding participants' prospective intention to use psycho-oncological support services ("Do you intend to use the in-house psycho-oncological support service in the next months?", answer options: yes, maybe, no), the recommendation by the dermatologist for psychological support as well as patients' real uptake (hospital record).
Patients' subjective experience and evaluation of modern technological examination | up to 24 months
  Study specific questions concerning the individuals' perceptions focusing the benefits by potentially improved sensitivity and specificity and possible disadvantages of the additional technology (3D TBP) in melanoma screening will be asked. The psychological impact of 3D TBP usage in melanoma screening and its effect on patients' cancer worry will be evaluated.

OTHER OUTCOMES:
Comparison of automated naevus counts from 3D total-body photography | Up to 3 years
  Comparison of automated naevus counts from 3D total-body photography generated by collegues in Australia
Impact of sun damage on diagnostic accuracy of DEXI algorithm in melanoma recognition | Up to 3 years
  Determination of the impact of sun damage on diagnostic accuracy of DEXI algorithm in melanoma recognition
Patient perception of AI utilisation in skin cancer screening via questionaire | Up to 3 years
  Including willingness to pay for 3D TBP
Comparison of the diagnostic accuracy of different algorithms by using ROC-AUC curves | Up to 3 years
  Investigating how different algorithms might change diagnostic accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Lara Valeska Maul, Dr. med., Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Goessinger EV, Niederfeilner JC, Cerminara S, Maul JT, Kostner L, Kunz M, Huber S, Koral E, Habermacher L, Sabato G, Tadic A, Zimmermann C, Navarini A, Maul LV. Patient and dermatologists' perspectives on augmented intelligence for melanoma screening: A prospective study. J Eur Acad Dermatol Venereol. 2024 Dec;38(12):2240-2249. doi: 10.1111/jdv.19905. Epub 2024 Feb 27. PMID 38411348
- [Derived] Goessinger EV, Cerminara SE, Mueller AM, Gottfrois P, Huber S, Amaral M, Wenz F, Kostner L, Weiss L, Kunz M, Maul JT, Wespi S, Broman E, Kaufmann S, Patpanathapillai V, Treyer I, Navarini AA, Maul LV. Consistency of convolutional neural networks in dermoscopic melanoma recognition: A prospective real-world study about the pitfalls of augmented intelligence. J Eur Acad Dermatol Venereol. 2024 May;38(5):945-953. doi: 10.1111/jdv.19777. Epub 2023 Dec 29. PMID 38158385
- [Derived] Cerminara SE, Cheng P, Kostner L, Huber S, Kunz M, Maul JT, Bohm JS, Dettwiler CF, Geser A, Jakopovic C, Stoffel LM, Peter JK, Levesque M, Navarini AA, Maul LV. Diagnostic performance of augmented intelligence with 2D and 3D total body photography and convolutional neural networks in a high-risk population for melanoma under real-world conditions: A new era of skin cancer screening? Eur J Cancer. 2023 Sep;190:112954. doi: 10.1016/j.ejca.2023.112954. Epub 2023 Jun 24. PMID 37453242